CLINICAL TRIAL: NCT02420782
Title: A Phase 1 Combined Single and Multiple Ascending Oral Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ASP6282 in Healthy Nonelderly and Elderly Male and Female Subjects, Including a Food Effect Cohort and Drug-drug Interaction Cohort With Itraconazole
Brief Title: First-in-human: Single Ascending Dose, Food Effect, Drug-drug Interaction, Multiple Ascending Dose, Proof of Pharmacology
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 6282-CL-0001; 2015-000093-35 (EudraCT Number)
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics; ASP6282; Pharmacodynamics; Drug-drug interaction; Midazolam; Safety and tolerability; Healthy volunteers; Itraconazole
MeSH Terms: interventions — Itraconazole; Pilocarpine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (10):
- ASP6282 single ascending dose (fasted) (Experimental): Part 1
  Interventions: Drug: ASP6282
- Placebo single ascending dose (fasted) (Placebo Comparator): Part 1
  Interventions: Drug: Placebo
- ASP6282 single dose (fed) (Experimental): Part 1
  Interventions: Drug: ASP6282
- Placebo single dose (fed) (Placebo Comparator): Part 1
  Interventions: Drug: Placebo
- ASP6282 single dose (fasted) (Experimental): Part 1 Period 1
  Interventions: Drug: ASP6282
- Itraconazole multiple dose and ASP6282 single dose (fasted) (Experimental): Part 1 Period 2
  Interventions: Drug: ASP6282; Drug: Itraconazole
- ASP6282 multiple ascending dose (nonelderly and elderly) (Experimental): Part 2. Germany only: once daily dosing, optional twice daily dosing. Midazolam dosing elderly only, exploratory for DDI purpose
  Interventions: Drug: ASP6282; Drug: Midazolam
- Placebo multiple ascending dose (nonelderly and elderly) (Placebo Comparator): Part 2. Germany only: once daily dosing, optional twice daily dosing
  Interventions: Drug: Placebo
- ASP6282 and pilocarpine (Experimental): Part 3
  Interventions: Drug: ASP6282; Drug: Pilocarpine
- Placebo and pilocarpine (Other): Part 3
  Interventions: Drug: Pilocarpine; Drug: Placebo

INTERVENTIONS:
Drug: ASP6282 — oral
  Arms: ASP6282 and pilocarpine; ASP6282 multiple ascending dose (nonelderly and elderly); ASP6282 single ascending dose (fasted); ASP6282 single dose (fasted); ASP6282 single dose (fed); Itraconazole multiple dose and ASP6282 single dose (fasted)
Drug: Itraconazole — oral
  Arms: Itraconazole multiple dose and ASP6282 single dose (fasted)
Drug: Pilocarpine — oral
  Arms: ASP6282 and pilocarpine; Placebo and pilocarpine
Drug: Placebo — oral
  Arms: Placebo and pilocarpine; Placebo multiple ascending dose (nonelderly and elderly); Placebo single ascending dose (fasted); Placebo single dose (fed)
Drug: Midazolam — oral
  Other Names: Versed
  Arms: ASP6282 multiple ascending dose (nonelderly and elderly)

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics (PK) and pharmacodynamics (PD) of single and multiple ascending oral doses of ASP6282 in healthy male and female subjects. 1 cohort (elderly) receives also a midazolam dosing.

This study will also explore the effect of itraconazole (another drug) on the PK of ASP6282, as well as to evaluate the safety and tolerability of ASP6282 alone and in combination with itraconazole in healthy male and female subjects.

Also, this study is to evaluate the PD and PK effects of single oral doses of ASP6282 on pilocarpine-induced salivation and pupil diameter in healthy nonelderly male and female subjects.

DETAILED DESCRIPTION:
This study consists of three parts. Part 1 is Single Ascending Dose Including Food Effect and Drug-drug Interaction (DDI) with Itraconazole. There will be a washout between treatment period 1 and 2 in the DDI arm of Part 1; Part 2 is a Multiple Ascending Dose (MAD); Part 3, with a treatment period 1, 2 and 3 is Proof of Pharmacology. There will be a washout between each treatment period

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index (BMI) range of 18.5 to 30.0 kg/m2, inclusive. The subject weighs at least 50 kg [screening].
* Female subject must not donate ova starting at screening and throughout the clinical study period, and for 28 days after the final study drug administration.
* Male subject and his female spouse/partners who are of childbearing potential must be using highly effective contraception consisting of 2 forms of birth control (1 of which must be a barrier method) starting at screening and continue throughout the clinical study period, and for 90 days after the final study drug administration.
* Male subject must not donate sperm starting at screening and throughout the clinical study period, and for 90 days after last study drug administration.
* Subject agrees not to participate in another interventional study while participating in the present clinical study, defined as signing the informed consent form until completion of the last study visit.

Germany only:

* Female subject must either:

  * Be of nonchildbearing potential:

    1. Postmenopausal (defined as at least 1 year without any menses) prior to screening, or,
    2. Documented surgically sterile.
  * Or, if of childbearing potential:

    1. Agree not to try to become pregnant during the clinical study and for 90 days after the final study drug administration,
    2. Must have a negative serum pregnancy test at day -1, and
    3. If heterosexually active, agree to consistently use a form of highly effective birth control in combination with a barrier method starting at screening and continuing throughout the clinical study period, and for 90 days after the final study drug administration.
    4. Or agree to stay abstinent, if abstinence is the preferred and usual lifestyle of the subject, starting at screening and continuing throughout the clinical study period and for 90 days after the final study drug administration.
* Female subject must agree not to breastfeed starting at screening and throughout the clinical study period, and for 90 days after the final study drug administration.
* Female subject must not donate ova starting at screening and throughout the clinical study period, and for 90 days after the final study drug administration.

Exclusion Criteria:

* Female subject who has been pregnant within 6 months prior to screening assessment or breastfeeding within 3 months prior to screening.
* Subject has a known or suspected hypersensitivity to ASP6282, itraconazole (part 1 - DDI only) or pilocarpine (part 3 - Proof of pharmacology (PoP) only) or any components of the formulations used.
* Subject uses a CYP3A4 metabolized substrate that can prolong the QT interval, e.g., astemizole, bepridil, cisapride, dofetilide, levacetylmethadol (levomethadyl), mizolastine, pimozide, quinidine, sertindole and terfenadine.
* Subject uses any of the following medication: atorvastatin, lovastatin and simvastatin, triazolam, midazolam, ergot alkaloids such as dihydroergotamine, ergometrine (ergonovine), ergotamine and methylergometrine (methylergonovine), eletriptan and nisodipine.
* Subject with evidence of ventricular dysfunction such as congestive heart failure or a history of congestive heart failure.
* Subject has clinically significant, cardiorenal disease, asthma and/or any other disease at risk for cholinergic agonists.
* Subject has a condition of the eye which could be affected by the intake of pilocarpine (e.g., acute iritis) (part 3 - PoP only).
* Subject has any of the liver chemistry tests (Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), alkaline phosphatase (ALP), gamma glutamyl transferase (GGT), Total bilirubin (TBL) above the Upper limit of normal (ULN)). In such a case, the assessment may be repeated once on Day -1 (in part 1 - DDI: treatment period 1 only).
* Subject has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Subject has chronic bronchitis and/or chronic obstructive pulmonary disease, or known or suspected cholelithiasis or biliary tract disease, or peptic ulceration or cognitive or psychiatric disturbances, or renal or hepatic insufficiency, or narrow-angle glaucoma.
* Subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection) or fungal (noncutaneous) infection within 1 week prior to admission to the clinical unit on Day -1.
* Subject has any clinically significant abnormality following the investigator's review of the physical examination, ECG and clinical study protocol-defined clinical laboratory tests at screening or day -1.
* Subject has a mean pulse < 40 or > 90 bpm; mean systolic blood pressure (SBP) > 140 mmHg; mean diastolic blood pressure (DBP) > 90 mmHg (vital signs measurements taken in triplicate after subject has been resting in supine position for 5 minutes; pulse will be measured automatically) on admission to the clinical unit on Day -1. If the mean blood pressure exceeds the limits above, 1 additional triplicate can be taken.
* Subject has a mean corrected QT interval using Fridericia's formula (QTcF) > 430 ms (for male subjects) and > 450 ms (for female subjects) at screening. If the mean QTcF exceeds the limits above, 1 additional triplicate ECG can be taken at screening.
* Subject uses any prescribed or nonprescribed drugs (including vitamins, natural and herbal remedies, e.g., St. John's wort) in the 2 weeks prior to first study drug administration, except for occasional use of paracetamol (up to 2 g/day) (all parts) and except for use of contraceptives or hormone replacement therapy (except for part 1- DDI).
* Subject has a history of smoking within 6 months prior to first study drug administration on day 1.
* Subject has a history of drinking > 21 units of alcohol/week for male subjects or > 14 units of alcohol/week for female subjects (1 unit = 10 g pure alcohol = 250 mL of beer [5%] or 35 mL of spirits [35%] or 100 mL of wine [12%]) within 3 months prior to admission to the clinical unit on Day -1.
* Subject has consumed grapefruit/Seville oranges, grapefruit-containing products or Seville orange-containing products within 72 hours prior to admission to the clinical unit on Day -1.
* Subject uses any inducer of metabolism (e.g., barbiturates, rifampin) within 1 month prior to admission to the clinical unit on Day -1.
* Subject uses any drugs of abuse within 3 months prior to admission to the clinical unit on Day -1.
* Subject had significant blood loss, donated 1 unit (500 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to admission to the clinical unit on Day -1.
* Subject has a positive serology test for hepatitis B surface antigen (HBsAg), hepatitis A virus antibodies (anti-HAV) (immunoglobulin M [IgM]), hepatitis C virus antibodies (anti-HCV), or antibodies to human immunodeficiency virus type 1 (HIV-1) and/or type 2 (HIV-2) at screening.
* Subject participated in any clinical study or has been treated with any investigational drugs within 90 days prior to screening.

Germany only:

* Subject has a mean pulse < 50 or > 90 bpm; mean systolic blood pressure (SBP) > 140 mmHg; mean diastolic blood pressure (DBP) > 90 mmHg (vital signs measurements taken in triplicate after subject has been resting in supine position for 5 minutes; pulse will be measured automatically) on admission to the clinical unit on day -1. (For elderly subjects the following criteria apply: SBP > 160 mmHg and DBP > 100 mmHg). If the mean blood pressure exceeds the limits above, 1 additional triplicate can be taken.
* Subject has a mean corrected QT interval using Fridericia's formula (QTcF) > 430 ms (for male subjects) and > 450 ms (for female subjects) at day -1. If the mean QTcF exceeds the limits above, 1 additional triplicate ECG can be taken at day -1.
* Subject has a positive serology test for hepatitis B surface antigen (HBsAg), hepatitis B core antibodies, hepatitis A virus antibodies (anti-HAV) (immunoglobulin M [IgM]), hepatitis C virus antibodies (anti-HCV), or antibodies to human immunodeficiency virus type 1 (HIV-1) and/or type 2 (HIV-2) at screening.
* Subject is unable to communicate, read and understand German, or has any other condition which, in the investigator's opinion, makes the subject unsuitable for clinical study participation.
* Subject is a vulnerable subject (e.g., subject kept in detention).
* Subject has a known or suspected hypersensitivity to ASP6282, itraconazole (part 1 - DDI only), pilocarpine (part 3 - PoP only) or midazolam (part 2 - elderly cohort only) or any components of the formulations used.
* Subject uses any prescribed or nonprescribed drugs (including vitamins, natural and herbal remedies, e.g., St. John's wort) in the 2 weeks prior to first study drug administration, except for occasional use of paracetamol (up to 2 g/day) (all parts) and except for use of hormone replacement therapy (except for part 1 - DDI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2015-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by adverse events | Part 1: up to 10 days; Part 2 up to 18 days
Safety as assessed by vital signs | Part 1: up to 10 days; Part 2 up to 18 days
  Vital signs include: blood pressure, pulse rate and body temperature
Safety as assessed by safety laboratory tests | Part 1: up to 10 days; Part 2 up to 18 days
  Laboratory tests include: hematology, biochemistry and urinalysis
Safety as assessed by electrocardiogram (ECG) measurements (Part 1) | From screening to end of study visit (ESV) (up to day 10)
  ECG measurements include routine ECG
Safety as assessed by continuous cardiac monitoring (Part 1) | From day 1 up to day 5
  12- lead ECG continuous cardiac monitoring, real-time cardiac monitoring (telemetry), cardiac troponin
Safety as assessed by electrocardiogram (ECG) measurements (Part 2) | From screening to ESV (Up to day 18)
  ECG measurements include routine 12- lead ECG, cardiac troponin
Safety as assessed by continuous electrocardiogram (ECG) measurements (Part 2) | From screening up to day 15
  Twelve lead continuous cardiac monitoring, cardiac troponin
Safety as assessed by the Orthostatic challenge test (OCT) (Part 1) | From day -1 up to day 5
  Blood pressure measurement
Pharmacodynamic parameter salivary secretion at specified timepoints (Part 3) | Day 1, each treatment period
  Measured (mg/min) salivary secretion at specific timepoints
Pharmacodynamic parameter salivary secretion AUEsal (Part 3) | Day 1, each treatment period
  Area under the effect curve salivary secretion (AUEsal)
Pharmacodynamic parameter salivary secretion Emax,sal (Part 3) | Day 1, each treatment period
  Maximum pharmacodynamic effect salivary secretion (Emax,sal)
Pharmacodynamic parameter salivary secretion tmax,sal (Part 3) | Day 1, each treatment period
  Time at maximum concentration salivary secretion (tmax,sal)

SECONDARY OUTCOMES:
Pharmacokinetics profile of ASP6282 (plasma): AUCinf, AUClast, Cmax, CL/F, tlag, tmax, t½, Vz/F (Part 1) | Day 1 up to Day 5, each treatment period
  Area under the concentration-time curve from the time of dosing extrapolated to time infinity (AUCinf); Area under the concentration-time curve from the time of dosing to the last measurable concentration (AUClast); Maximum concentration (Cmax); Apparent total systemic clearance after extravascular dosing (CL/F); Time prior to the time corresponding to the first measurable (nonzero) concentration (tlag);Time at maximum concentration (tmax); Terminal elimination half-life (t½); Apparent volume of distribution during the terminal elimination phase after extravascular dosing (Vz/F)
Pharmacokinetics profile of ASP6282 (urine): Aelast, Aelast%, Aeinf, Aeinf%, CLR (Part 1) | Day 1 up to Day 4, each treatment period
  Cumulative amount of study drug excreted into urine from time of dosing up to the collection time of the last measurable concentration (Aelast); Percentage of study drug dose excreted into urine from time of dosing up to the collection time of the last measurable concentration (Aelast%); Cumulative amount of study drug excreted into urine from time of dosing extrapolated to time infinity (Aeinf); Percentage of study drug dose excreted into urine from time of dosing extrapolated to time infinity (Aeinf%); Renal clearance (CLR)
Pharmacokinetic parameter of Itraconazole (plasma) Ctrough (Part 1) | Day 1 up to Day 5, each treatment period
  DDI arm only. Concentration immediately prior to dosing at multiple dosing (Ctrough)
Pharmacokinetics profile of ASP6282 (plasma): AUC24, tlag, AUCtau, CL/F, PTR, Rac(AUC), Cmax, tmax, t½, Vz/F (Part 2) | Day 1 up to Day 20
  Area under the concentration-time curve from the time of dosing to 24 hours postdose (AUC24); Area under the concentration-time curve from the time of dosing to the start of the next dosing interval (AUCtau); Peak trough ratio (PTR), Accumulation ratio calculated using the area under the concentration-time curve (Rac(AUC))
Pharmacokinetics profile of ASP6282 (urine): Aetau, Aetau%, CLR (Part 2) | Day 14
  Percentage of study drug dose excreted into urine over the time interval between consecutive dosing (Aetau%)
Pharmacokinetics profile of ASP6282 (plasma): AUC6, AUCinf, AUClast, Cmax, CL/F, tlag, tmax, t½, Vz/F (Part 3) | Day 1 up to Day 5, per treatment period
  Area under the concentration-time curve from the time of dosing to 6 hours Postdose (AUC6)
Pharmacokinetics profile of Pilocarpine (plasma): AUC6, Cmax, tmax (Part 3) | Day 1, per treatment period
Pharmacodynamic profile pupil diameter pupS, AUEpupS, Emax,pupS, tmax,pupS, (Part 1, Part 2) | Part 1: Day 1; Part 2: Day -1 and Day 14
  Part 1: exclusive DDI arm. Pupil diameter, scotopic lighting condition (pupS); Area under the effect curve pupil diameter, scotopic lighting condition (AUEpupS); Maximum pharmacodynamic effect pupil diameter, scotopic lighting condition (Emax,pupS), Time at maximum concentration pupil diameter, scotopic lighting condition (tmax,pupS)
Pharmacodynamic profile salivary secretion AUEsal, Emax,sal, tmax,sal (Part 1, Part 2) | Part 1: Screening and Day 1; Part 2: Day -1 and Day 14
  Part 1: exclusive DDI arm
Pharmacodynamic profile of Bond and Lader VAS (Part 1, Part 2) | Part 1: Day 1; Part 2: Day -1 and Day 14
  Visual analogue scale (VAS)
Safety profile assessed by nature, frequency and severity of adverse events, vital signs, safety laboratory tests and 12 lead ECG (Part 3) | Screening, Day -1 and ESV (Day 10)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Clinical Pharmacology & Exploratory Development (CPED)
Locations (2):
- Site DE49001, Berlin, Germany
- Site GB44001, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided